CLINICAL TRIAL: NCT02752490
Title: The Comparative Effectiveness of Liberal Versus Restricted Maternal Administration of Oxygen During Labor: a Controlled Before and After Study
Brief Title: The Comparative Effectiveness of Liberal Versus Restricted Maternal Administration of Oxygen During Labor
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Nanaama Ankumah Bentum, Clinical Fellow PGY 6, The University of Texas Health Science Center, Houston
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HSC-MS-16-0142
Record Dates: First submitted 2016-04-20; First posted 2016-04-27 (Estimated); Results first posted 2018-03-02 (Actual); Last update posted 2020-10-12 (Actual); Status verified 2020-10

CONDITIONS: Maternal Oxygen Use in Labor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Liberal use of maternal oxygen (Active Comparator): Administration of maternal oxygen, 100% FiO2 at 10L/min via nonrebreather face mask with any category 2 tracing as defined by the American Congress of Obstetrics and Gynecology (ACOG) at the discretion of the primary nurse or physician
  Interventions: Drug: Liberal use of maternal oxygen
- Indicated use of maternal oxygen (Experimental): Administration of maternal oxygen, 100% fraction of inspired oxygen (FiO2) at 10 liters/min via nonrebreather face mask only in the setting of a category 2 tracing with recurrent late fetal heart rate decelerations, prolonged fetal deceleration, fetal tachycardia, or minimal to absent fetal heart rate variability lasting 30 minutes or greater. Maternal oxygen is discontinued once these conditions have resolved and may be readministered if they recur.
  Interventions: Drug: Indicated use of maternal oxygen

INTERVENTIONS:
Drug: Liberal use of maternal oxygen — Administration of maternal oxygen, 100% FiO2 at 10L/min via nonrebreather face mask with any category 2 tracing as defined by ACOG10 at the discretion of the primary nurse or physician
  Arms: Liberal use of maternal oxygen
Drug: Indicated use of maternal oxygen — Administration of maternal oxygen, 100% FiO2 at 10L/min via nonrebreather face mask only in the setting of a category 2 tracing with recurrent late fetal heart rate decelerations, prolonged fetal deceleration, fetal tachycardia, or minimal to absent fetal heart rate variability lasting 30 minutes or greater. Maternal oxygen is discontinued once these conditions have resolved and may be readministered if they recur.
  Arms: Indicated use of maternal oxygen

SUMMARY:
The objective of this study is to determine if a strategy of indicated compared to liberal oxygen administration in labor decreases the rate of cesarean delivery. The hypothesis is that women who undergo a strategy of indicated compared to liberal oxygen administration in labor will have lower rate of cesarean delivery and fetal acidemia at birth.

DETAILED DESCRIPTION:
This is a single-site before and after study comparing the strategy of liberal versus indicated use of maternal oxygen in the first and second stages of labor in the setting of a category 2 fetal heart rate tracing (FHR) tracing, as defined by American Congress of Obstetrics and Gynecology (ACOG) and National Institute of Child Health and Human Development (NICHD) guidelines. All patients who are at term and are undergoing labor at Memorial Hermann Hospital in Houston, Texas during the time frame of the study will be included in the study. The study will be conducted over 18 weeks. It will involve two 8 week time periods during which all patients will under either a strategy of liberal administration of oxygen use (current practice) in the "before" portion of the study and indicated administration of oxygen in the "after" portion of the study (new practice). There will be a transition period where training, education, and audit + feedback will be done to prepare for a strategy of indicated administration of oxygen.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women with singleton gestation between 37 weeks 0 days to 42 weeks 0 days gestation who present to labor and delivery at Memorial Hermann Hospital in Houston, TX for planned labor attempt.

Exclusion Criteria:

* Lethal fetal anomaly defined as anomaly in which the fetus is unlikely to survive or the neonate is not expected to survive to initial hospital discharge
* Antepartum or intrapartum fetal demise
* Preexisting maternal conditions requiring oxygen for maternal indication, including but not limited to: Asthma that has required intubation or hospitalization in the past or currently requiring steroids (either inhaled or oral); Chronic obstructive pulmonary disease; Chronic bronchitis; Congestive heart failure/peripartum cardiomyopathy; Pneumonia; Pulmonary edema; Pulmonary embolus

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 844 (Actual)
Dates: Start 2016-04; Primary Completion 2016-07-31 (Actual); Study Completion 2016-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nana-Ama E Ankumah, MD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- Children's Memorial Hermann Hospital, Houston, Texas, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Liberal Use of Maternal Oxygen | Indicated Use of Maternal Oxygen
Started | 409 | 435
Completed | 409 | 435
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Liberal Use of Maternal Oxygen | Indicated Use of Maternal Oxygen | Total
Number analyzed (Participants) | 409 | 435 | 844
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.7 (5.6) | 27.7 (5.6) | 27.7 (5.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 409 | 435 | 844
  Male | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 409 | 435 | 844

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Delivered by Cesarean
Time Frame: at time of birth
Measure: Count of Participants; unit: Participants
Arm/Group | Liberal Use of Maternal Oxygen | Indicated Use of Maternal Oxygen
Number analyzed (Participants) | 409 | 435
Participants | 83 | 75

2. Secondary Outcome: Number of Participants With Umbilical Artery pH (Potential Hydrogen) < 7.10 at Birth
Time Frame: at time of birth
Population: For this outcome measure, the number of participants analyzed is not equal to the number of participants who started or completed the study because each participant's provider determines whether umbilical artery pH is analyzed, and thus, umbilical artery pH is not collected for every participant in the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Liberal Use of Maternal Oxygen | Indicated Use of Maternal Oxygen
Number analyzed (Participants) | 227 | 243
Participants | 7 | 12

3. Secondary Outcome: Number of Participants Who Delivered by Cesarean for Non-reassuring Fetal Status
Time Frame: at time of birth
Measure: Count of Participants; unit: Participants
Arm/Group | Liberal Use of Maternal Oxygen | Indicated Use of Maternal Oxygen
Number analyzed (Participants) | 83 | 75
Participants | 37 | 39

4. Secondary Outcome: Number of Participants Whose Infants Had an Apgar Score < 7 at 5 Minutes
Description: The Apgar score is based on a total score of 1 to 10. The higher the score, the better the baby is doing after birth. A score of 7, 8, or 9 is normal and is a sign that the newborn is in good health. A score of 10 is very unusual, since almost all newborns lose 1 point for blue hands and feet, which is normal for after birth.
Time Frame: 5 minutes after birth
Measure: Count of Participants; unit: Participants
Arm/Group | Liberal Use of Maternal Oxygen | Indicated Use of Maternal Oxygen
Number analyzed (Participants) | 409 | 435
Participants | 4 | 13

5. Secondary Outcome: Number of Participants Whose Infants Were Admitted to the Neonatal Intensive Care Unit (NICU)
Time Frame: from time of birth to discharge from hospital (an average of 2-4 days)
Measure: Count of Participants; unit: Participants
Arm/Group | Liberal Use of Maternal Oxygen | Indicated Use of Maternal Oxygen
Number analyzed (Participants) | 409 | 435
Participants | 38 | 42

6. Secondary Outcome: Total Duration of Maternal Oxygen Use
Time Frame: during labor
Population: For this outcome measure, the number of participants analyzed is not equal to the number of participants who started or completed the study because not all participants received oxygen. All who received oxygen were analyzed for this measure.
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | Liberal Use of Maternal Oxygen | Indicated Use of Maternal Oxygen
Number analyzed (Participants) | 217 | 216
minutes | 89 [42 to 172] | 87 [36 to 152]

7. Secondary Outcome: Number of Participants Who Received Intrauterine Resuscitation Other Than Administration of Maternal Oxygen
Description: "Intrauterine resuscitation" includes administration of terbutaline, amnioinfusion, cessation of oxytocin, and intravenous (IV) fluid boluses. In this measure, the number of participants who received any of these 5 procedures will be reported in aggregate as the "number of participants who received intrauterine resuscitation other than administration of maternal oxygen."
Time Frame: during labor
Measure: Count of Participants; unit: Participants
Arm/Group | Liberal Use of Maternal Oxygen | Indicated Use of Maternal Oxygen
Number analyzed (Participants) | 409 | 435
Participants
  Administration of intravenous fluid bolus | 240 | 236
  Cessation of oxytocin | 121 | 118
  Amnioinfusion | 13 | 11
  Administration of terbutaline | 18 | 23

8. Secondary Outcome: Number of Participants With Clinical Chorioamnionitis
Time Frame: during labor
Measure: Count of Participants; unit: Participants
Arm/Group | Liberal Use of Maternal Oxygen | Indicated Use of Maternal Oxygen
Number analyzed (Participants) | 409 | 435
Participants | 16 | 14

ADVERSE EVENTS:
Arm/Group | Liberal Use of Maternal Oxygen | Indicated Use of Maternal Oxygen
Serious Adverse Events (participants affected / at risk) | 0/409 | 0/435
Other Adverse Events (participants affected / at risk) | 0/409 | 0/435

LIMITATIONS AND CAVEATS:
This was a non-randomized trial, and was performed in a single institution, which may reduce its generalizability.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes